CLINICAL TRIAL: NCT01295216
Title: Mobile Health to Prevent Progression of Pre-hypertension in Latin American Urban Settings
Brief Title: Use of Mobile Technology to Prevent Progression of Pre-hypertension in Latin American Urban Settings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No significant change for the primary objective at 12 months
Sponsor: Institute of Nutrition of Central America and Panama (Other)
Collaborators: Institute for Clinical Effectiveness and Health Policy (Other); Universidad Peruana Cayetano Heredia (Other); RAND (Other)
Responsible Party: Principal Investigator, Manuel Ramirez-Zea, Head, INCAP Comprehensive Center for the Prevention of Chronic Diseases, Institute of Nutrition of Central America and Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HHSN268200900028C
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Hypertension; Prehypertension
Keywords: prehypertension; blood pressure; mobile technology; Latin America; behavioral change; healthy lifestyles; mHealth
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Pre-hypertensive subjects who receive mHealth support for 12 months
  Interventions: Behavioral: Mobile technology to promote lifestyle modification
- Control (No Intervention): Individuals who receive the usual primary health care

INTERVENTIONS:
Behavioral: Mobile technology to promote lifestyle modification — Effects of an intervention using mobile health (mHealth) technology, including short message services (SMS) and one-to-one telephone calls, to promote lifestyle modification focused on reducing blood pressure among participants
  Arms: Intervention

SUMMARY:
Nearly half of the adult population in Latin American urban settings has abnormally high blood pressure. Although half of these subjects with high blood pressure are still in the pre-hypertensive stage (systolic blood pressure values in the 120-139 mmHg range or diastolic blood pressure in the 80-89 mmHg range), the rate of progression to hypertension is high (10-20% per year), according to studies done in other settings. The main objective of this proposal is to evaluate the effectiveness of an affordable and sustainable primary health care intervention to reduce blood pressure and prevent progression from pre-hypertensive status to hypertension in individuals at poor urban clinics in Argentina, Guatemala, and Peru. Our primary hypotheses are that pre-hypertensive subjects who receive mHealth (mobile health) support for 12 months (intervention group) will have lower blood pressure compared to individuals who receive the usual primary health care (control group); and that pre-hypertensive subjects will maintain lower blood pressure six months after receiving mHealth support. The investigators will determine the effects of an intervention using mHealth technology, including short message services (SMS) and one-to-one telephone calls, to promote lifestyle modification focused on reducing blood pressure among participants. The intervention also aims to help participants become better informed, motivated, and encouraged to practice self-management of their own health; to improve patient satisfaction levels; provide tailored targeted interventions; and to improve patient-provider relationships. The proposal is designed as a proof-of-concept intervention in three Latin American countries that encompass a wide range of environments and health care settings. A total of 212 subjects (30-60 years old) per country will be recruited in primary health clinics and randomized to study groups. Blood pressure, anthropometry, and behavioral risk factors (physical activity, diet, stress, alcohol and tobacco use) will be measured at baseline and at months 6 and 12 during the intervention, and six months after the end of the intervention. The investigators will also evaluate feasibility, acceptability, cost-effectiveness, and process implementation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure values in the 120-139 mmHg range or diastolic blood pressure in the 80-89 mmHg range
* No current anti-hypertensive medication
* Own a personal cellular phone

Exclusion Criteria:

* Previous diagnosis/treatment hypertension
* Illiteracy
* Another household member already in the study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 637 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Institute for Clinical Effectiveness and Health Policy, Buenos Aires, Argentina
- Insitute of Nutrition of Central America and Panama, Guatemala City, Guatemala
- Universidad Peruana Cayetano Heredia, Lima, Peru

REFERENCES:
- [Derived] Bernabe-Ortiz A, Pauschardt J, Diez-Canseco F, Miranda JJ. Sustainability of mHealth Effects on Cardiometabolic Risk Factors: Five-Year Results of a Randomized Clinical Trial. J Med Internet Res. 2020 Apr 21;22(4):e14595. doi: 10.2196/14595. PMID 32314970
- [Derived] Carrillo-Larco RM, Jiwani SS, Diez-Canseco F, Kanter R, Beratarrechea A, Irazola V, Ramirez-Zea M, Rubinstein A, Martinez H, Miranda JJ; GISMAL Group. Implementation Tells Us More Beyond Pooled Estimates: Secondary Analysis of a Multicountry mHealth Trial to Reduce Blood Pressure. JMIR Mhealth Uhealth. 2018 Nov 1;6(11):e10226. doi: 10.2196/10226. PMID 30389646
- [Derived] Rubinstein A, Miranda JJ, Beratarrechea A, Diez-Canseco F, Kanter R, Gutierrez L, Bernabe-Ortiz A, Irazola V, Fernandez A, Letona P, Martinez H, Ramirez-Zea M; GISMAL group. Effectiveness of an mHealth intervention to improve the cardiometabolic profile of people with prehypertension in low-resource urban settings in Latin America: a randomised controlled trial. Lancet Diabetes Endocrinol. 2016 Jan;4(1):52-63. doi: 10.1016/S2213-8587(15)00381-2. Epub 2015 Dec 1. PMID 26653067

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 316 | 321
Completed | 266 | 287
Not Completed | 50 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 316 | 321 | 637
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (8.4) | 43.2 (8.4) | 43.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 173 | 342
  Male | 147 | 148 | 295
Region of Enrollment [Number; unit: participants]
  Argentina | 104 | 108 | 212
  Guatemala | 105 | 108 | 213
  Peru | 107 | 105 | 212

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure at 6, 12, and 18 Months
Description: A reduction in systolic and diastolic blood pressure is expected as early as 6 months of intervention and it is expected that this reduction is maintained or even continue to decrease over time
Time Frame: Baseline, 6, 12, and 18 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 316 | 321
mmHg
  Systolic blood pressure, 12 months | -5.23 [-6.45 to -3.86] | -4.89 [-6.19 to -3.59]
  Diastolic blood pressure, 12 months | -2.34 [-3.28 to -1.41] | -2.32 [-3.27 to -1.37]
  Systolic blood pressure, 6 months | -5.13 [-6.40 to -3.86] | -4.01 [-5.21 to -2.81]
  Diastolic blood pressure, 6 months | -1.82 [-2.71 to -0.93] | -1.36 [-2.20 to -0.52]
  Systolic blood pressure, 18 months | NA [NA to NA] — No data were collected at the 18-month time point | NA [NA to NA] — No data were collected at the 18-month time point
  Diastolic blood pressure, 18 months | NA [NA to NA] — No data were collected at the 18-month time point | NA [NA to NA] — No data were collected at the 18-month time point
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority or Other; Mean Difference (Net) = -0.37, 95% CI 2-sided [-2.15 to 1.40] — Systolic blood pressure at 12 months
Statistical Analysis 2: Comparison: Intervention vs Control; Test type: Superiority or Other; Mean Difference (Net) = 0.01, 95% CI 2-sided [-1.29 to 1.32] — Diastolic blood pressure for 12 months

2. Secondary Outcome: Change From Baseline in Food Intake at 12 Months
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: Servings/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 316 | 321
Servings/day
  Fruit&Veg intake (servings/day) | 0.35 [0.14 to 0.57] | 0.10 [-0.06 to 0.26]
  High-sodium food intake (servings/day) | -0.41 [-0.55 to -0.27] | -0.36 [-0.49 to -0.23]
  High-fat & sugar food intake (servings/day) | -1.86 [-2.27 to -1.45] | -1.16 [-1.54 to -0.78]

3. Secondary Outcome: Change From Baseline in Body Weight at 12 Months
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 316 | 321
kg | -0.18 [-0.66 to 0.29] | 0.48 [0.08 to 0.90]

4. Secondary Outcome: Change From Baseline in Body Mass Index at 12 Months
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: kg/m2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 316 | 321
kg/m2 | -0.10 [-0.27 to 0.08] | 0.19 [0.03 to 0.35]

5. Secondary Outcome: Change From Baseline in Waist Circumference at 12 Months
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Intervention | Control
Number analyzed (Participants) | 316 | 321
cm | 0.03 [-0.71 to 0.77] | 0.61 [-0.06 to 1.27]

6. Secondary Outcome: Change From Baseline in Physical Activity at 12 Months
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: MET/min/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 316 | 321
MET/min/week | -88.3 [-318.8 to 142.2] | -20.7 [-228.0 to 186.6]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/316 | 0/321
Other Adverse Events (participants affected / at risk) | 0/316 | 0/321

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No